CLINICAL TRIAL: NCT03568643
Title: Azithromycin as Adjunctive Therapy for Uncomplicated Severe Acute Malnutrition:
Brief Title: Azithromycin for Uncomplicated Severe Acute Malnutrition in Burkina Faso (Pilot)
Acronym: SAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-25274; 1R21HD100932-01A1 (NIH)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Uncomplicated Severe Acute Malnutrition
MeSH Terms: interventions — Azithromycin; Amoxicillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Experimental): children in this arm will receive one dose of azithromycin
  Interventions: Drug: Azithromycin
- Amoxicillin (Active Comparator): Children in this arm will receive a 7 day course of amoxicillin (standard of care)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Azithromycin — Children enrolled in the trial and randomized to azithromycin will receive a single directly observed dose of oral azithromycin at 20 mg/kg up to the maximum adult dose of 1 g. Oral azithromycin will be administered at the time of enrollment. Enrolled children will also receive RUTF.
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Amoxicillin — Children enrolled in the trial and randomized to azithromycin will receive a 7-day course of oral amoxcillin given in twice-daily doses of 50-100 mg/kg, per the Burkina Faso guidelines for the management of severe acute malnutrition. The first dose will be administered at the time of enrollment and the remaining dose will be administered by the caregiver at home. Enrolled children will also receive RUTF.
  Arms: Amoxicillin

SUMMARY:
This pilot study is a randomized controlled trial designed to test the effect of the administration of adjunctive azithromycin in conjunction with standard outpatient treatment for uncomplicated severe acute malnutrition (SAM) in children aged 6-59 months. Children presenting to nutritional programs in Burkina Faso who meet eligibility criteria will be randomized to a single dose of oral azithromycin or a 7-day course of amoxicillin (standard of care) upon admission into the program. All enrolled children will receive ready-to-use therapeutic foods (RUTF). Enrolled children will be followed at each weekly clinic follow-up visit up to 8 weeks following admission. Data on anthropometric indicators, vital status, and adverse events will be collected during follow-up. Nutritional recovery over the 8-week study period will be compared by arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months
* WHZ <-3 SD or MUAC <115 mm
* No nutritional edema
* Able and willing to participate in full 8-week study
* Has not been admitted to a nutritional program for the treatment of SAM in the 3 preceeding months
* No antibiotic use in past 7 days
* No clinical complications requiring inpatient treatment (except for routine admission for children <6 months)
* No congenital abnormality or chronic debilitating illness that would lead to predictable growth faltering or reduce likelihood of SAM treatment benefit (such as cerebral palsy, Down syndrome, congenital heart disease, cleft lip/palate, etc)
* No allergy to macrolides/azalides
* Sufficient appetite according to a feeding test with ready-to-use therapeutic food (RUTF)
* Appropriate consent from at least one parent or guardian

Exclusion Criteria:

* Age <6 months or >59 months
* WHZ ≥-3 SD or MUAC ≥115 mm
* Nutritional edema
* Not able or willing to participate in full 8-week study
* Admission to a nutritional program for the treatment of SAM in the 3 preceeding months
* Antibiotic use in past 7 days
* Clinical complications requiring inpatient treatment
* Congenital abnormality or chronic debilitating illness that would lead to predictable growth faltering or reduce likelihood of SAM treatment benefit (such as cerebral palsy, Down syndrome, congenital heart disease, cleft lip/palate, etc)
* Allergy to macrolides/azalides
* Insufficient appetite according to a feeding test with ready-to-use therapeutic food (RUTF)
* Parent or guardian refuses to provide consent

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Oldenburg, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de Recherche en santé de nouna, Nouna, Boucle du Mouhoun, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldenburg CE, Hinterwirth A, Dah C, Millogo O, Coulibaly B, Ouedraogo M, Sie A, Chen C, Zhong L, Ruder K, Lebas E, Nyatigo F, Arnold BF, O'Brien KS, Doan T. Gut Microbiome among Children with Uncomplicated Severe Acute Malnutrition in a Randomized Controlled Trial of Azithromycin versus Amoxicillin. Am J Trop Med Hyg. 2022 Dec 12;108(1):206-211. doi: 10.4269/ajtmh.22-0381. Print 2023 Jan 11. PMID 36509053
- [Derived] Oldenburg CE, Hinterwirth A, Ourohire M, Dah C, Ouedraogo M, Sie A, Boudo V, Chen C, Ruder K, Zhong L, Lebas E, Nyatigo F, Arnold BF, O'Brien KS, Doan T. Gut Resistome after Antibiotics among Children with Uncomplicated Severe Acute Malnutrition: A Randomized Controlled Trial. Am J Trop Med Hyg. 2022 Jun 13;107(1):59-64. doi: 10.4269/ajtmh.22-0007. Print 2022 Jul 13. PMID 35895362
- [Derived] Sie A, Dah C, Ourohire M, Ouedraogo M, Boudo V, Arzika AM, Lebas E, Nyatigo F, Arnold BF, O'Brien KS, Oldenburg CE. Azithromycin versus Amoxicillin and Malarial Parasitemia among Children with Uncomplicated Severe Acute Malnutrition: A Randomized Controlled Trial. Am J Trop Med Hyg. 2021 Sep 27;106(1):351-355. doi: 10.4269/ajtmh.21-0595. PMID 34583344
- [Derived] O'Brien KS, Sie A, Dah C, Ourohire M, Arzika AM, Boudo V, Lebas E, Godwin WW, Arnold BF, Oldenburg CE. Azithromycin for uncomplicated severe acute malnutrition: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Apr 20;7(1):97. doi: 10.1186/s40814-021-00836-w. PMID 33879263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin | Amoxicillin
Started | 161 | 140
Completed | 161 | 140
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Amoxicillin | Total
Number analyzed (Participants) | 161 | 140 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 161 | 140 | 301
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 16.9 (8.4) | 16.5 (8.2) | 16.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 77 | 169
  Male | 69 | 63 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 161 | 140 | 301
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 161 | 140 | 301
Curently breastfeeding [Number; unit: Participants] | 108 | 104 | 212
Exclusively breastfeeding [Number; unit: Participants] | 10 | 11 | 21
Number of children under 5 in the household [Mean (Standard Deviation); unit: Children] | 2 (1.7) | 1.9 (1.5) | 1.9 (1.6)
Mother's age [Mean (Standard Deviation); unit: years] | 26 (6.2) | 26.2 (6) | 26.1 (6.1)
Weight [Mean (Standard Deviation); unit: Kg] | 6.8 (1.3) | 6.6 (1.3) | 6.7 (1.3)
Height [Mean (Standard Deviation); unit: cm] | 72.2 (6.6) | 71.6 (6.6) | 71.9 (6.6)
MUAC (Middle Upper Arm Circumference) [Mean (Standard Deviation); unit: cm] — Mid-Upper Arm Circumference (MUAC) is the circumference of the left upper arm, measured at the mid-point between the tip of the shoulder and the tip of the elbow (olecranon process and the acromium). MUAC is used for the assessment of nutritional status.
  MUAC less than 11.5cm is considered as severe malnutrition
  cm | 11.2 (0.4) | 11.2 (0.5) | 11.2 (0.5)
HAZ (Height for Age Z-score) [Mean (Standard Deviation); unit: Z score] — A z-score of 0 represents the population mean. The z-score will be positive if the data value lies above the mean, and negative if the data value lies below the mean
  The score was calculated using the 2006 World Health Organization's Child Growth Standards:
  Stunted is length/height-for-age below the -2 z-score line. Severely stunted is below the -3 z-score line
  Z score | -2.4 (1.5) | -2.5 (1.6) | -2.4 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain
Description: Weight will be measured at all follow-up time points and weight gain will be calculated at 8 weeks
Time Frame: 8 weeks
Population: All children who were followed up to 8 weeks. This analysis excludes 19 children who were lost to follow-up before 8 weeks.
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
g/kg/day | 1.8 (2.1) | 2.0 (2.2)

2. Secondary Outcome: Nutritional Recovery - Primary Definition
Description: Nutritional recovery is defined as, depending on admission criteria: weight-for-height/length is equal to or more than -2 Z-score and the child have had no oedema for at least 2 weeks, or the mid-upper-arm circumference is equal to or more than 125 mm and the child have had no oedema for at least 2 weeks.
  Anthropometric outcomes were defined according to the 2006 World Health Organization's Child Growth Standards:
  Stunted is length/height-for-age below the -2 z-score line. Severely stunted is below the -3 z-score line
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Participants | 56 | 48

3. Secondary Outcome: Nutritional Recovery - Secondary Definition
Description: Summarize the cumulative proportion recovered by arm. Children are considered recovered if they had mean upper arm circumference > 12.5 or weight-for-height/length > -2 for 2 consecutive measurements. Additionally, it includes children who had had mean upper arm circumference >12.5 or weight-for-height/length > -2 on their final measurement, regardless of whether they met these criteria on the previous visit.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Participants | 98 | 87

4. Secondary Outcome: Malaria
Description: Rapid diagnostic tests for malaria will be conducted at baseline and week 8 to determine malaria infection status.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Participants | 13 | 15

5. Secondary Outcome: Mortality
Description: Vital status will be assessed at all follow-up time points and mortality will be defined as death during the study period.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Participants | 2 | 1

6. Secondary Outcome: Length/Height-for-age Z-score (LAZ/HAZ)
Description: Height or length will be measured at all follow-up time points and height-for-age z-scores will be calculated.
  A z-score of 0 represents the population mean. The z-score will be positive if the data value lies above the mean, and negative if the data value lies below the mean.
  Anthropometric outcomes were defined according to the 2006 World Health Organization's Child Growth Standards:
  Stunted is length/height-for-age below the -2 z-score line. Severely stunted is below the -3 z-score line
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Z-score | -2.3 (1.5) | -2.37 (1.5)

7. Secondary Outcome: Mid-Upper Arm Circumference (MUAC)
Description: Mid-upper arm circumference will be measured at all follow-up time points
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
cm | 12.4 (0.8) | 12.3 (0.8)

8. Secondary Outcome: Weight-for-Age Z-scores (WAZ)
Description: Weight will be measured at all follow-up time points and weight-for-age z-scores will be calculated.
  A z-score of 0 represents the population mean. The z-score will be positive if the data value lies above the mean, and negative if the data value lies below the mean.
  Anthropometric outcomes were defined according to the 2006 World Health Organization's Child Growth Standards:
  Underweight is weight-for-age below the -2 z-score line. Severely underweight is below the -3 z-score line.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Z-score | -2.58 (1.1) | -2.65 (1.1)

9. Secondary Outcome: Weight-for-Height Z-score (WHZ)
Description: Weight and height, assessed at all follow-up time points, will be used to calculate weight-for-height z-scores.
  A z-score of 0 represents the population mean. The z-score will be positive if the data value lies above the mean, and negative if the data value lies below the mean.
  Anthropometric outcomes were defined according to the 2006 World Health Organization's Child Growth Standards:
  Overweight is weight-for-length/height above the 2 z-score line. Severely overweight; weight-for-length/height above the 3 z-score line
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 150 | 132
Z-score | -1.89 (1.2) | -1.95 (1.0)

10. Secondary Outcome: Intestinal Microbiome
Description: baseline and 8 week intestinal microbiome will be compared between the 2 arms alpha diversity using inverse Simpson's index and Shannon's index, expressed in effective number.
  The Shannon Diversity Index is a quantitative measure that reflects how many different bacterial species there are in a sample. The greater the index, the more diverse the gut microbiota. An index of 0 indicates a community that only has one species. A negative change indicates a decrease in diversity and a positive change indicates an increase in diversity.
  The Simpson's Diversity Index is a measure of diversity which takes into account the number of species present, as well as the relative abundance of each species. As species richness and evenness increase, so diversity increases. The value ranges between 0 and 1, where 1 represents infinite diversity and 0, no diversity.
Time Frame: Baseline, 8 weeks
Population: Children who had a rectal swab collected at baseline and at 8 weeks.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Azithromycin | Amoxicillin
Number analyzed (Participants) | 49 | 46
Index
  Baseline Simpson's Index | 4.0 (2.6) | 5.1 (3.5)
  Baseline Shannon's Index | 6.6 (4.4) | 8.3 (5.6)
  Week 8 Simpson's Index | 4.5 (2.8) | 5.3 (2.9)
  Week 8 Shannon's Index | 7.5 (4.6) | 9.1 (5.8)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Cumulative number of adverse event incidences over a period of 8 weeks.
Arm/Group | Azithromycin | Amoxicillin
All-Cause Mortality (participants affected / at risk) | 2/161 | 1/140
Serious Adverse Events (participants affected / at risk) | 41/161 | 43/140
Other Adverse Events (participants affected / at risk) | 106/161 | 100/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=161) | Amoxicillin (N=140)
Hospitalization (Surgical and medical procedures) | 2 (2) | 3 (4) — Hospitalized by 8 weeks
Clinic visit (Surgical and medical procedures) | 41 (59) | 42 (58) — Sought medical care by 8 weeks
Death (Cardiac disorders) | 2 (2) | 1 (1) — Death by week 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=161) | Amoxicillin (N=140)
fever (Infections and infestations) | 82 (131) | 80 (134)
Diarrhea (Gastrointestinal disorders) | 46 (62) | 44 (62)
Vomiting (Gastrointestinal disorders) | 33 (42) | 23 (33)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 6 (7)
skin rash (Skin and subcutaneous tissue disorders) | 7 (10) | 16 (22)
constipation (Gastrointestinal disorders) | 7 (8) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03568643/Prot_SAP_000.pdf